CLINICAL TRIAL: NCT01984463
Title: Impact of Epidural Morphine on the Incidence and Severity of Shoulder Pain Following Thoracotomy.
Brief Title: Impact of Epidural Morphine on Shoulder Pain Following Thoracotomy.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Increased incidence of respiratory depression in the morphine group
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13.203
Record Dates: First submitted 2013-11-04; First posted 2013-11-14 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Postoperative Pain; Shoulder Pain
Keywords: Postoperative pain; Shoulder pain; Thoracotomy
MeSH Terms: conditions — Pain, Postoperative; Shoulder Pain | interventions — Fentanyl; Morphine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fentanyl (Active Comparator): Patients will be randomized to receive by the epidural catheter a bolus dose of 100 mcg of fentanyl followed by an infusion of epidural bupivacaine 0.1% and fentanyl 2 mcg/mL.
  Interventions: Drug: Fentanyl
- Morphine (Experimental): Patients will be randomized to receive by the epidural catheter a bolus dose of 3 mg of morphine followed by an infusion of epidural bupivacaine 0.1% and morphine 50 mcg/mL.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Fentanyl — Patients will receive an epidural bolus dose of 100 mcg of fentanyl followed by an infusion of epidural bupivacaine 0.1% and fentanyl 2 mcg/mL continued postoperatively until the surgical drains are removed or for a maximum of five days.
  Other Names: Epidural fentanyl
  Arms: Fentanyl
Drug: Morphine — Patients will receive an epidural bolus dose of 3 mg of morphine followed by an infusion of epidural bupivacaine 0.1% and morphine 50 mcg/mL continued postoperatively until the surgical drains are removed or for a maximum of five days.
  Other Names: Epidural morphine
  Arms: Morphine

SUMMARY:
This study is designed to assess the impact of epidural morphine on:

* The incidence and severity of shoulder pain following a thoracotomy.
* The need for additional analgesics, such as opioids for the relief of shoulder pain.
* Its safety profile compared to epidural fentanyl following a thoracotomy.

The basic hypothesis of this study is that an infusion of epidural bupivacaine and morphine initiated after the induction of anesthesia and continued until 72 hours postoperatively will reduce the incidence and severity of shoulder pain following a thoracotomy when compared to an epidural infusion of bupivacaine and fentanyl.

DETAILED DESCRIPTION:
Despite adequate epidural analgesia, up to 97% of patients undergoing thoracotomy will experience ipsilateral shoulder pain. Although this pain is well recognized, its cause remains unclear. Several mechanisms have been suggested to explain this pain, including somatic and visceral as well as phrenic nerve nociception. The phrenic nerve arises from the third to the fifth cervical nerves and provides the sensory innervation for the mediastinal and diaphragmatic pleura and pericardium. Patients will complain of a constant, moderate to severe aching pain, in the posterior deltoid and in the suprascapular region, ipsilateral to the surgery. Different treatments have been used to alleviate post-thoracotomy shoulder pain, but few of these efforts have been proven effective and safe.

A mixture of epidural bupivacaine and fentanyl is considered the standard of care for post-thoracotomy analgesia in our center. The infusion is started after induction of anesthesia with a bolus dose followed with a continuous infusion and bolus doses as needed for the following days. To optimize the use of epidural analgesia after thoracotomy, it would seem well-advised to try to reach higher dermatomes. This could possibly be achieved by using a different opioid in combination with bupivacaine in the epidural infusion. Morphine could be an interesting agent in order to reach cervical spinous dermatomes probably involved in the genesis of post-thoracotomy shoulder pain.

Methods: The anesthetic technique and monitoring will be standardized. Prior to the induction of general anesthesia, a thoracic epidural catheter will be inserted under local anesthesia between the fourth and the eight spinous processes. Correct placement of the epidural will be assessed. A bolus dose of fentanyl 100 mcg or morphine 3 mg will be given by the epidural catheter as per randomization. The epidural infusion will be initiated at a rate of 0.1 mL/kg/hr before surgery and continued postoperatively until the surgical drains are removed or for a maximum of five days. To relieve thoracic pain, the epidural infusion rate will be adjusted up to a maximum of 12 mL/hr, with boluses of 0.05 mL/kg as needed. Hydromorphone will be used postoperatively as rescue analgesia for shoulder pain. All patients will receive standardised doses of acetaminophen for the first 48 hours following surgery.

On arrival in the recovery room, correct placement of the epidural will be reassessed. During the immediate postoperative period, the intensity of pain will be assessed using a Verbal Numeric Pain Scale (0-10). Pain will be assessed at 2,4,8,12 and 24 hours after surgery and daily thereafter, for a total duration of 4 postoperative days. Interference of pain with daily activities will be assessed using the Brief Pain Inventory (BPI) at 24 hours following surgery. Signs of neuropathic pain will be assessed using the Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) scale at 24 hours following surgery.

Side-effects attributable to analgesia will be recorded. Arterial blood samples will be collected every 8 hours for the first 24 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 75 years
* Scheduled for an elective thoracotomy
* Physical status 1-3

Exclusion Criteria:

* Contraindication to epidural analgesia (coagulopathy, sepsis or local infection at the site of injection, spinal deformity, previous major spinal thoracic surgery)
* A known allergy to local anesthetics, acetaminophen, fentanyl or morphine.
* Pre-existing shoulder pain ipsilateral to the surgery
* Pre-existing chronic pain
* Current use of opioids
* Recent history of alcohol or drug abuse.
* The inability to understand a verbal numerical pain scale (VNPS) despite previous instruction
* Severe renal insufficiency
* Patient refusal

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Intensity of pain using a Verbal Numeric Pain Scale (VNPS) | From arrival in the recovery room until 4 days after surgery or discharge from the hospital, the first to occur.

SECONDARY OUTCOMES:
Opioid consumption | From arrival in the recovery room until 4 days after surgery or discharge from the hospital, the first to occur.
Side-effects attributable to analgesia | From surgery until 4 days after surgery or discharge from the hospital, the first to occur.
Interference of pain with daily activities using the Brief Pain Inventory | 24 hours after surgery.
Signs of neuropathic pain using the Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) scale | 24 hours after surgery.
Impact of epidural morphine on gas exchange by measuring arterial blood gases | Every 8 hours for the first 24 hours following surgery.

CONTACTS AND LOCATIONS:
Overall Officials: François Girard, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada